CLINICAL TRIAL: NCT05162534
Title: Evaluation of Independent Clinical- Laboratory Predictors of Clinical Outcomes in Hospitalized Positive SARS-CoV2 Patients (Outcomes SARS-CoV2)
Brief Title: Independent Predictors on Clinical Outcomes in SARS-CoV2 Patients
Acronym: outcomes
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Collaborators: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Angelina Passaro, Professor, University Hospital of Ferrara
Other Study IDs: 520/2020/Oss/AOUFe
Record Dates: First submitted 2021-12-09; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: COVID-19 Patients
Keywords: COVID-19; SARS-CoV-2; mortality risk prediction
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients needing IoC: Patients needing IoC can be recognized by the acronym "IoCp"
  Interventions: Other: effect of COVID-19 exposure
- 30-day deceased patients: Patient died after a period of observation of 30 days are presented with the acronyms "30-ddp" (30-day deceased patients)
  Interventions: Other: effect of COVID-19 exposure
- did not undergo IoC: Patients did not undergo IoC, we chose the acronym "nIoCp".
  Interventions: Other: effect of COVID-19 exposure
- 30-day survived patients: Patient survived after a period of observation of 30 days are presented with the acronyms "30-dsp" (30-day survived patients)
  Interventions: Other: effect of COVID-19 exposure

INTERVENTIONS:
Other: effect of COVID-19 exposure — effect of COVID-19 exposure

SUMMARY:
The clinical spectrum of COVID-19 can be very heterogeneous: from mild flu-like symptoms, to the form with severe pulmonary impairment (dyspnoea, tachypnoea, PaO2 / FiO2 ratio below 300 at arterial blood gas sampling, pulmonary infiltrates covering more than 50% of the respiratory surface); up to 5% of patients tend to rapidly develop acute respiratory distress syndrome (ARDS) with or without acute cardiac damage, underlying a phase of systemic hyperinflammation (cytokine storm) that may result in shock, multi-organ failure and death

DETAILED DESCRIPTION:
AIM OF THE STUDY The purpose of the study is to evaluate the existence of prognostic indices of the disease starting from the anamnestic, clinical and laboratory data of the patients belonging to the medical departments of the S. Anna Hospital in Cona (Fe), partially dedicated to COVID-19 patients.

OBJECTIVES

Primary:

• Evaluation of prognostic indices determining the need for intensification of care, in-hospital and 30-day mortality in hospitalized patients tested positive for SARS-CoV-2 infection

Secondary:

* Evaluation of prognostic indices determining the need for intensification of care, in-hospital and 30-day mortality in hospitalized patients with SARS-CoV-2 infection
* Evaluation of organ damage by collecting the main organ-specific damage indices (TnI HS, CPK, LDH, ALT, isoamylase, creatinine) associated with SARS-CoV-2 infection.

METHODS The retrospective observational study will be conducted from March 2020 to May 2020 in the medical departments of Internal Medicine, Pulmonology and in the Intensive Care Units of the S.Anna Hospital in Cona (Fe), Italy.

Participants will be recruited from patients belonging to the facilities of the semi-intensive and intensive medical departments of the health company of Ferrara's province.

Anamnestic, clinical and laboratory data will be collected from the medical records of hospitalized patients. All patients of both sexes, over the age of 18 admitted to the above medical wards, with confirmed positivity to the nasopharyngeal swab for SARS-CoV-2 will be recruited.

INCLUSION CRITERIA

* Males and Females older than 18 years
* Infection by SARS-CoV-2 confirmed with at least one positive naso-pharyngeal swab
* Patient hospitalized for COVID-19 in the medical ward, semi-intensive and intensive

EXCLUSION CRITERIA

* Patients younger than 18 years
* Doubtful or unconfirmed swab detection of SARS-CoV-2 The study did not require the collection of written or verbal consent: for its drafting, in fact, only anamnestic and laboratory data were obtained, without needing to collect biological samples.

We have decided to enroll in the study the patients hospitalized for COVID-19 in the departments of internal medicine, pulmonology and in the intensive care units of the province of Ferrara.

Clinical surveillance: Evaluation of anamnestic and laboratory data extrapolated from the medical records of individual patients.

ELIGIBILITY:
INCLUSION CRITERIA Males and Females older than 18 years Infection by SARS-CoV-2 confirmed with at least one positive naso-pharyngeal swab Patient hospitalized for COVID-19 in the medical ward, semi-intensive and intensive EXCLUSION CRITERIA Patients younger than 18 years Doubtful or unconfirmed swab detection of SARS-CoV-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We evaluated the differences between subjects in terms of the three major COVID-19 outcomes (1. IoC=intensification of care, meant as the need for non-invasive mechanical ventilation or for endotracheal intubation; 2. in-hospital death; 3. 30-day death).
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | Observation during hospitalisation or 30 days after diagnosis
  Evaluation of prognostic indices determining the need for intensification of care, in-hospital and 30-day mortality in hospitalized patients tested positive for SARS-CoV-2 infection

SECONDARY OUTCOMES:
Secondary Outcome | Observation during hospitalisation or 30 days after diagnosis
  Evaluation of prognostic indices determining the need for intensification of care, in-hospital and 30-day mortality in hospitalized patients with SARS-CoV-2 infection
Secondary Outcome 2 | Observation during hospitalisation or 30 days after diagnosis
  Evaluation of organ damage by collecting the main organ-specific damage indices (TnI HS, CPK, LDH, ALT, isoamylase, creatinine) associated with SARS-CoV-2 infection.

CONTACTS AND LOCATIONS:
Overall Officials: Angelina Passaro, MD, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- University Hospital of Ferrara Arcispedale Sant'Anna, Ferrara, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madjid M, Safavi-Naeini P, Solomon SD, Vardeny O. Potential Effects of Coronaviruses on the Cardiovascular System: A Review. JAMA Cardiol. 2020 Jul 1;5(7):831-840. doi: 10.1001/jamacardio.2020.1286. PMID 32219363
- [Background] Godeau D, Petit A, Richard I, Roquelaure Y, Descatha A. Return-to-work, disabilities and occupational health in the age of COVID-19. Scand J Work Environ Health. 2021 Jul 1;47(5):408-409. doi: 10.5271/sjweh.3960. Epub 2021 May 18. No abstract available. PMID 34003294
- [Result] Song Z, Xu Y, Bao L, Zhang L, Yu P, Qu Y, Zhu H, Zhao W, Han Y, Qin C. From SARS to MERS, Thrusting Coronaviruses into the Spotlight. Viruses. 2019 Jan 14;11(1):59. doi: 10.3390/v11010059. PMID 30646565
- [Result] Zhang JJ, Dong X, Cao YY, Yuan YD, Yang YB, Yan YQ, Akdis CA, Gao YD. Clinical characteristics of 140 patients infected with SARS-CoV-2 in Wuhan, China. Allergy. 2020 Jul;75(7):1730-1741. doi: 10.1111/all.14238. Epub 2020 Feb 27. PMID 32077115
- [Result] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Result] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Result] Li B, Yang J, Zhao F, Zhi L, Wang X, Liu L, Bi Z, Zhao Y. Prevalence and impact of cardiovascular metabolic diseases on COVID-19 in China. Clin Res Cardiol. 2020 May;109(5):531-538. doi: 10.1007/s00392-020-01626-9. Epub 2020 Mar 11. PMID 32161990
- [Result] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Result] Zhang W, Zhao Y, Zhang F, Wang Q, Li T, Liu Z, Wang J, Qin Y, Zhang X, Yan X, Zeng X, Zhang S. The use of anti-inflammatory drugs in the treatment of people with severe coronavirus disease 2019 (COVID-19): The Perspectives of clinical immunologists from China. Clin Immunol. 2020 May;214:108393. doi: 10.1016/j.clim.2020.108393. Epub 2020 Mar 25. PMID 32222466
- [Result] Goyal P, Choi JJ, Pinheiro LC, Schenck EJ, Chen R, Jabri A, Satlin MJ, Campion TR Jr, Nahid M, Ringel JB, Hoffman KL, Alshak MN, Li HA, Wehmeyer GT, Rajan M, Reshetnyak E, Hupert N, Horn EM, Martinez FJ, Gulick RM, Safford MM. Clinical Characteristics of Covid-19 in New York City. N Engl J Med. 2020 Jun 11;382(24):2372-2374. doi: 10.1056/NEJMc2010419. Epub 2020 Apr 17. No abstract available. PMID 32302078
- [Result] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385